Smart Television and Exercise Promotion for Independent Living Facilities (STEP4Life)

Data Analysis Plan

NCT03001778

8/19/2014

## **Step for Life Data Analysis Plan**

Usability testing will be recorded, transcribed, coded, and analyzed with constant comparative and phenomenological approaches, using Atlas.ti™. We will identify problems that impact >10% of ILF users. For a 95% chance of detection (log(1-.95)/log(1-.10)), usability testing of 28 ILF OAs is needed. With non-ILF users, we will have a 95% chance of detection for problems impacting >15% (n=20)